CLINICAL TRIAL: NCT03358849
Title: Phase 1 Clinical Trial to Evaluate the Safety of Allogeneic NK Cell ("SMT-NK") Cell Therapy in Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-1165
Record Dates: First submitted 2017-11-21; First posted 2017-12-02 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Advanced Biliary Tract Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental)
  Interventions: Biological: Natural killer cell

INTERVENTIONS:
Biological: Natural killer cell — Patients who received natural killer cell injection
  Other Names: SMT-NK cell

SUMMARY:
Cholangiocarcinoma refers to bile duct cancer (bile duct cancer) and gallbladder cancer that develop in the gallbladder. According to the data from National Cancer Information Center in 2013, the incidence of cancer in Korea is 5,283, which corresponds to about 2.3% of all cancers and the 5-year survival rate is 30% And most of the long-term survival is due to early detection by screening, and advanced carcinoma is a refractory carcinoma with a 5-year survival rate of less than 5%. In addition to the standard anticancer drugs, alternative anticancer drugs and targeted therapies have been developed to provide a variety of treatment modalities. However, the development of cell therapy drugs for cancer, such as cancers, has not been developed in Korea. .

Natural killer cells (NK cells) are innate lymphocyte cells with cytotoxic activity. Unlike T cells and B cells, which have antigen-specific receptors, NK cells express various innate immunoreceptors on the cell surface, thereby enabling selective recognition of cancer cells And recognizes cancer cells, it is a cytotoxic cell that can immediately remove cancer cells without any other activation process. In addition, natural killer cells also interact with dendritic cells or T cells directly or indirectly to regulate the immune response, thereby inhibiting the development and metastasis of cancer cells and effectively removing cancer stem cells important for cancer recurrence It has many advantages in the development of anti-cancer immunotherapy.

DETAILED DESCRIPTION:
Cholangiocarcinoma refers to bile duct cancer (bile duct cancer) and gallbladder cancer that develop in the gallbladder. According to the data from National Cancer Information Center in 2013, the incidence of cancer in Korea is 5,283, which corresponds to about 2.3% of all cancers and the 5-year survival rate is 30% And most of the long-term survival is due to early detection by screening, and advanced carcinoma is a refractory carcinoma with a 5-year survival rate of less than 5%. In addition to the standard anticancer drugs, alternative anticancer drugs and targeted therapies have been developed to provide a variety of treatment modalities. However, the development of cell therapy drugs for cancer, such as cancers, has not been developed in Korea. .

Although surgical resection is mandatory for curettage of the biliary tract, 40 ~ 50% of all patients are able to undergo radical resection. In general, the incidence of mid / lower bile duct cancer is high and the upper bile duct cancer is relatively low. The surgical resection of the tumor depends on the location of the tumor. The curative surgery of the biliary cancer is very complicated and time-consuming. The anatomical structures of the biliary and vascular system are variable and it is difficult to accurately determine the extent of the tumor invasion before surgery or even during surgery there is also a great deal of risk. Especially in the case of hepatic portal biliary duct (upper bile duct cancer), it is difficult to judge whether surgical resection is feasible, and there are many cases where resection is difficult at the time of operation or discovery. Gallbladder cancer also has a poor prognosis. Early cancer can be cured by surgery, but progressive cancer has a poor prognosis and overall survival rate is similar to that of biliary cancer. Because it occurs in the biliary tract with bile duct cancer, the clinical method and characteristics of the cancer cells are similar, and the same method is used for the treatment and the chemotherapy.

However, since there is no standard for the selection of second-line chemotherapy after gemcitabine treatment, the development of an alternative therapeutic agent is urgently required have.

Natural killer cells (NK cells) are innate lymphocyte cells with cytotoxic activity. Unlike T cells and B cells, which have antigen-specific receptors, NK cells express various innate immunoreceptors on the cell surface, thereby enabling selective recognition of cancer cells And recognizes cancer cells, it is a cytotoxic cell that can immediately remove cancer cells without any other activation process. In addition, natural killer cells also interact with dendritic cells or T cells directly or indirectly to regulate the immune response, thereby inhibiting the development and metastasis of cancer cells and effectively removing cancer stem cells important for cancer recurrence It has many advantages in the development of anti-cancer immunotherapy.

Therefore, various clinical studies have been conducted to treat cancer using natural killer cells worldwide, including in Korea, and therapeutic clinical results are shown for various cancers. The clinical application of natural killer cells is carried out by culturing natural killer cells isolated from blood of patient, patient's family or even from other people's blood and injecting them into patients. It is also possible to expect the effect as a combination therapy with chemotherapy alone or by eliminating the cancer cells in the patient's body while improving the immunity of the patient by improving the immunity of the patient.

However, despite this, the clinical application of natural killer cells in Korea is limited to only a few cancers, including hematologic and hepatocellular carcinoma.

Carcinoid cancer (biliary cancer, gallbladder cancer) is a rare carcinoma with around 3,500 cases per year in Korea. In the majority of cases, the rate of relying entirely on chemotherapy is more than 50%, and the response rate of Gemcitabine based on the first chemotherapy is about 30%. Other alternative therapies that do not lead to cancer are natural killer cells that need to be tested for safety and efficacy in existing drugs.

In Korea, the clinical application of natural killer cells is limited to only a few cancers, including hematologic and hepatocellular carcinomas. Carcinoid cancer (biliary cancer, gallbladder cancer) is a rare carcinoma with around 3,500 cases per year in Korea. In the majority of cases, the rate of relying entirely on chemotherapy is more than 50%, and the response rate of Gemcitabine based on the first chemotherapy is about 30%. Other alternative therapies that do not lead to cancer are natural killer cells that need to be tested for safety and efficacy in existing drugs.

ELIGIBILITY:
Inclusion Criteria:

* patients with pathologically proven biliary tract cancer (gallbladder cancer, cholangiocarcinoma),
* patients with refractory disease after chemotherapy and/or patients who have difficulty with chemotherapy due to side effects of chemotherapy
* 18y≤age≤75y
* ECOG performance status (ECOG-PS) ≤2
* Patients who meet the following conditions; 1)ANC ≥ 1,500/μL, 2) Hemoglobin) ≥ 10 g/dL, 3) PLT > 100,000/ μL, 4) Serum BUN & Creatinine ≤ 1.5 x ULN, 5) AST & ALT ≤ 2.5 x ULN, 6) Bilirubin ≤ 3mg/L
* Informed consent

Exclusion Criteria:

* Immune deficiency or autoimmune disease that can be exacerbated by immunotherapy
* Pregnancy
* Patients who have a history of other malignancies except skin cancer, local prostate cancer or cervical intraepithelial neoplasm within 5 years before the start of this study
* Serious allergic history, psychological disease
* Breast feeding or Patients planning pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 1 week after NK cell injection
  Adverse event and drug related toxicity will be checked every week by the investigator's monitoring.
Dose limiting toxicity | 2 weeks after NK cell injection
  Adverse event and drug related toxicity will be checked every week by the investigator's monitoring.
Dose limiting toxicity | 3 weeks after NK cell injection
  Adverse event and drug related toxicity will be checked every week by the investigator's monitoring.
Dose limiting toxicity | 4 weeks after NK cell injection
  Adverse event and drug related toxicity will be checked every week by the investigator's monitoring.
Maximum Tolerated Dose | 1 week after NK cell injection
  Adverse event and drug related toxicity will be checked every week by the investigator's monitoring.
Maximum Tolerated Dose | 2 weeks after NK cell injection
  Adverse event and drug related toxicity will be checked every week by the investigator's monitoring.
Maximum Tolerated Dose | 3 weeks after NK cell injection
  Adverse event and drug related toxicity will be checked every week by the investigator's monitoring.
Maximum Tolerated Dose | 4 weeks after NK cell injection
  Adverse event and drug related toxicity will be checked every week by the investigator's monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No